CLINICAL TRIAL: NCT01241110
Title: Phase 4 Study of Azitromicin in the Treatment of PID
Brief Title: To Compare Ofloxacin With Azitromycin for Pelvic Inflammatory Disease (PID) Treatment
Acronym: CTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guilan University of Medical Sciences (Other)
Responsible Party: fariba mirblook, GUMS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ClinicalTrials.gov; R01DA013131 (NIH)
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-10

CONDITIONS: Pelvic Inflammatory Disease
Keywords: PID, Ofloxacin, Azitromicine, Metronidazole
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- azitromicin,PID treatment,ofluxacin (Active Comparator)
  Interventions: Drug: Ofloxacin group A, Azitromycin group B; Drug: azitromycin

INTERVENTIONS:
Drug: Ofloxacin group A, Azitromycin group B — Group A (treated by Ofloxacin 400 mg. + Metronidazole 500mg) and Group B (a single dose of oral Azitromicine 1gr + Metronidazole 500mg) for 10 days, were compared in terms of side effects and efficacy.
  Other Names: azitromicin, ofluxacin
Drug: azitromycin — azitromicin vs ofluxacin
  Other Names: azitromicin; ofluxacin

SUMMARY:
Objective: To compare two oral treatments: Ofloxacin + Metronidazole, and Azitromycin +Metronidazole in outpatients with Pelvic Inflammatory Disease.

Materials and Methods: Two hundred patients divided to two groups( A , B). Group A (treated by Ofloxacin 400 mg. + Metronidazole 500mg) and Group B (a single dose of oral Azitromicine 1gr + Metronidazole 500mg) for 10 days, were compared in terms of side effects and efficacy

DETAILED DESCRIPTION:
Two hundred patients divided to two groups( A , B). Group A (treated by Ofloxacin 400 mg. + Metronidazole 500mg) and Group B (a single dose of oral Azitromicine 1gr + Metronidazole 500mg) for 10 days, were compared in terms of side effects and efficacy

ELIGIBILITY:
Inclusion Criteria:Eligibility criteria were having three out of five following symptoms: a-lower abdominal pain, b-vaginal discharges, c- adnexal tenderness, d-cervical motion tenderness (CMT), e-cervisitis.

-

Exclusion Criteria:Excluding criteria were as follows: a-unmarried women, b-pregnant women, c-women with infection during menstruation, d- history of abortion or miscarriage during the last month, e-underlying diseases such as diabetes, f-used antibiotics in the last month, or allergy to the antibiotics used in the study, g-history of Pelvic Inflammatory Disease within the last year, and h- suspicion of being multi partner.

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
to compare two oral antibiotic protocols in terms of side effects and efficacy. | Jan 2010- Aug 2010
  side effects- and efficacy

SECONDARY OUTCOMES:
single oral dose of Azitromicine could be the drug of choice in the outpatient treatment of Pelvic Inflammatory Disease | Jan 2010- Aug 2010
  compliance and cost

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Mirblook, MD, Principal Investigator — Guilan University of Medical Sciences
Locations (1):
- Alzahra Maternity Hospital, Rasht, Gilan Province, Iran